CLINICAL TRIAL: NCT02819934
Title: A Phase I Study to Investigate the Absorption, Metabolism, and Excretion of KD101 in Male Subjects
Brief Title: A Phase I Study to Investigate the ADME of KD101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Howard Lee, MD,PhD, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KD101_hAME
Record Dates: First submitted 2016-05-30; First posted 2016-06-30 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

ARMS (1):
- Arm1 (Experimental): experimental group
  Interventions: Drug: KD101

INTERVENTIONS:
Drug: KD101 — after 10 min KD101 administered, 14C KD101 3.52ug/1ml administrated. both of them will be administrate for oral

SUMMARY:
A Phase I Study to Investigate the Absorption, Metabolism, and Excretion of KD101 in Male Subjects

DETAILED DESCRIPTION:
A Phase I Study to Investigate the Absorption, Metabolism, and Excretion of KD101 in Male Subjects

ELIGIBILITY:
Inclusion Criteria:

* Are able to provide written informed consent
* The subject is a healthy Korean aged 20 to 55 years, inclusive.
* The subject weighs at least 55 and has a body mass index (BMI)over 27

Exclusion Criteria:

* Subjects with evidence or a history of clinically significant pulmonary, cardiovascular, hepatic, endocrine, hematological, neurologic or psychiatric diseases.
* Subjects with evidence of gastrointestinal disease which can affect the absorption of drug.
* Subjects with a history of drug abuse or a positive result in the urine drug screening for drug abuse
* Subjects who have taken any prescribed medicine or herbal medicine within 2 weeks before the first administration of the investigational product, any non-prescribed medicine or vitamin supplement within 1 week prior the first administration of the investigational product (if all other conditions are satisfied, subjects may be eligible for the trial as judged by the investigator.)
* Subjects who have donated a unit of whole blood within 30 days or who have participated in any other clinical trial within 60 days prior the first administration of the investigational product
* Subject who have history of allergy.
* Subject who can not continue proper contraception method during study period.
* Subjects who consume more than 21 units of alcohol per week (1 unit = 10 g of pure alcohol) or who are unable to abstain from drinking during the PK/PD testing period
* Subjects who are unable to abstain from smoking during the PK/PD testing period
* Subjects who are unable to abstain from grapefruit or caffeine containing food 1 day prior the first administration of the investigational product
* Subjects judged not eligible for the study after reviewing the clinical laboratory results or other reasons by the investigator.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2016-06-06 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Total radioactivity at feces,urine,blood to measure total recovery rate | 13day
  radioactivity in nCi